CLINICAL TRIAL: NCT00217061
Title: The Statin Choice Decision Aid and Its Effects on Statin Decisions in Patients With Type 2 Diabetes Mellitus. A Clustered Randomized Trial
Brief Title: Effect of a Decision Aid About Statin Use in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 38-05
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Diabetes Mellitus; Dyslipidemia; Hypercholesterolemia; Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus; Dyslipidemias; Hypercholesterolemia; Cardiovascular Diseases

INTERVENTIONS:
Device: Decision Aid Statin Choice

SUMMARY:
Background- Statins are a safe and effective therapy to reduce cardiovascular risk in patients with type 2 diabetes; however some patients are not prescribed statins, others do not take it even after being prescribed, and others stop therapy prematurely. Lack of knowledge or misinformation about statins may be responsible for inadequate statin use.

Objective- To test the hypothesis that a formal, structured decision aid could correct deficiencies in the current decision-making process, increase statin use, and improve outcomes in patients with type 2 diabetes.

Methods - The investigators will develop a decision aid called STATIN CHOICE and will pilot its efficacy in a blinded randomized controlled trial enrolling 98 type 2 diabetes patients.

Outcomes- Primary outcomes: adherence to the decision to use or not to use statins three months after using STATIN CHOICE. Secondary outcomes: acceptability of STATIN CHOICE, knowledge about options, satisfaction with decisions, decisional conflict, encounter duration, and quality of life.

Expected results- The investigators anticipate that this work will yield an effective and innovative decision aid for statin use in type 2 diabetes patients. STATIN CHOICE, along with a detailed users manual, will be directly applicable in clinical practice. Data and experience from this project will inform the planning and conduct of a randomized multicenter trial of the effectiveness of STATIN CHOICE in diverse practice settings.

Significance- Patient participation in decision-making resulting in informed treatment decisions, as proposed in this study, will likely lead to improved quality of decision-making, more appropriate use of statins, and improved patient outcomes.

ELIGIBILITY:
Adult patients with type 2 diabetes attending a referral diabetes clinic, who are taking or not taking statins, and give consent to participate. Excluded were patients who had sensory or mental impairments or language barriers that preclude them from using the intervention and therefore participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98
Dates: Start 2005-04; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Adherence to the decision to use or not to use statins

SECONDARY OUTCOMES:
Decisional conflict
Knowledge and understanding of risk
Quality of life (generic and disease specific)
Anxiety state
Trust in clinician

CONTACTS AND LOCATIONS:
Overall Officials: Victor M. Montori, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Wyatt KD, Branda ME, Inselman JW, Ting HH, Hess EP, Montori VM, LeBlanc A. Genders of patients and clinicians and their effect on shared decision making: a participant-level meta-analysis. BMC Med Inform Decis Mak. 2014 Sep 2;14:81. doi: 10.1186/1472-6947-14-81. PMID 25179289
- [Derived] Weymiller AJ, Montori VM, Jones LA, Gafni A, Guyatt GH, Bryant SC, Christianson TJ, Mullan RJ, Smith SA. Helping patients with type 2 diabetes mellitus make treatment decisions: statin choice randomized trial. Arch Intern Med. 2007 May 28;167(10):1076-82. doi: 10.1001/archinte.167.10.1076. PMID 17533211